CLINICAL TRIAL: NCT05512507
Title: Development of Sanomechanics® Rehabilitative Technology for Normalizing Contact Pressure in Painful Joints by Activating the Newly Discovered Floating Skeleton System.
Brief Title: Sanomechanics® Rehabilitative Technology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: PolyOrth International (Industry)
Responsible Party: Sponsor
Other Study IDs: POI 052022
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Physical Therapy Program — Physical Therapy Program

SUMMARY:
Rehabilitative Sanomechanics Method (RSM) of exercise designed to restore normal subperiosteal transmission of in-joint pressures and normalizing contact pressures on cartilages, will reduce pain in the affected joints and improve locomotor function.

DETAILED DESCRIPTION:
Specific Aim 1: In a clinical trial with subjects reporting arthritic knee pain, demonstrate that the Sanomechanics method of exercise, focused on restoring normal subperiosteal transmission of in-joint pressures, will reduce pain. Using the validated WOMAC questionnaire as a Patient- Reported Outcome (PRO) tool, the associated primary endpoint is that 80% of patients will report a reduction in pain at the end of the 3-month study based on the 5-point categorical WOMAC pain scale.

Specific Aim 2: To demonstrate that Sanomechanics will improve normal synergy in gait by mitigating compensatory gait strategy, which one develops to avoid unbearable pain in the joint. The associated co-primary endpoint is that 80% of patients will experience an increase in stance knee flexion angle. The secondary endpoint is that the 80% of patients will report a lowered WOMAC function score based on 5-point categorical WOMAC scale (lower score corresponds to better self-reported function) after the three-month study.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral knee pain with WOMAC score 6-9.
* Knee pain, aching or stiffness on most days in the past month and definite radiographic osteoarthritis in the index knee.
* Morning stiffness >30 min.
* Age: 40-75 years of age.
* More pain in the morning compared to evening.
* English speakers.
* Have daily access to an email address and a computer with Internet
* Allowed to be on prescription or non-prescription medicine for pain during the course of the study.

Exclusion Criteria:

* Inability to communicate in English
* Lower limb injury, surgery, or intra-articular injection in the past 6-months
* Current pregnancy
* Have a pacemaker or other internal medical device
* Cancer not in remission
* Gout
* History of stroke affecting lower limb
* Major trauma
* Gross knee instability on exam
* Lumbar radiculopathy affecting symptomatic limb
* KL radiographic score 4
* Morphological indications (bone-on-bone contact) for joint replacement

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study intends to enroll diversified patient population diagnosed with unilateral osteoarthritis of the knee
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The WOMAC self-reported pain score . | 90 days
  80% of patients will report a reduction in pain at the end of the 3-month study based on the 5-point categorical WOMAC pain scale.
The WOMAC self-reported function score | 90 days
  80% of patients will report a lowered WOMAC function score based on 5-point categorical WOMAC scale (lower score corresponds to better self-reported function) after the three-month study.

IPD SHARING:
Plan to Share IPD: No